CLINICAL TRIAL: NCT00121355
Title: An Open-Label, Multi-Center, Prospective Cross-Over Study of Preference and Safety of NovoFine® Autocover(TM) Needles Compared to BD Safety Glide (TM) Syringes in the Hospital Setting
Brief Title: Novofine Autocover Safety Needle Versus BD Safety Glide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MS241-1674
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Healthcare Professionals; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: safety glide
Device: autocover needle

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to examine whether nurses prefer to use the NovoFine® Autocover Needle or the BD Safety Glide (TM) Syringe (only) in a hospital setting. The number of needle stick injuries will also be evaluated and whether these hospital nurses prefer the safety features of the NovoFine® Autocover Needle versus those of the BD Safety Glide (TM) Syringe. The identified hospital nurses will evaluate the two types of needles during standard administration of insulin to patients being treated for diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Hospital nurses with prior injection training without an infectious blood borne disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Plainsboro, New Jersey, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com